CLINICAL TRIAL: NCT05340114
Title: Summative Usability Study of CEREBO® in Traumatic Brain Injury Patients to Determine Ease of Use, Ease of Learning and Satisfaction
Brief Title: Usability Study of CEREBO® - A Novel Non-invasive Intracranial Bleed Detector
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bioscan Research Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: BR/CV/2021/001; CTRI/2022/04/041634 (Registry Identifier: Clinical Trials Registry - India (ICMR-NIMS))
Record Dates: First submitted 2022-04-15; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Traumatic Brain Injury; Intracranial Hemorrhages
Keywords: Ease of Use; Ease of Learning; Satisfaction
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hemorrhages; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects examined by the operations with CEREBO® (Experimental): CEREBO® - A portable non-invasive device to detect intracranial haemorrhage Frequency - The operator will scan at least 10 patients Duration - 40 seconds per subject No adverse effect or contraindications
  Interventions: Device: CEREBO®

INTERVENTIONS:
Device: CEREBO® — Near-infrared based point-of-care portable intracranial hematoma detector

SUMMARY:
Traumatic Brain Injury (TBI) is the leading cause of death and disability across the globe. Time from injury to treatment is the most critical factor that determines the patient's recovery. Mild TBI with no apparent symptoms are often left undiagnosed, thus delaying the treatment and hence recovery. CEREBO® is a non-invasive, rapid, near-infrared based, point-of-care device that can detect an intracranial bleed at an early stage.

DETAILED DESCRIPTION:
This prospective study determines the usability of CEREBO® to detect the intracranial hematoma. The operators will receive a training session before the study and will be evaluated at the end of the study through a survey questionnaire for ease of use, ease of learning and satisfaction. Each operator will examine at least 10 subjects with CEREBO®.

ELIGIBILITY:
Inclusion Criteria:

Operators -

Medical health professionals >18 years of age with a valid medical license to practice medicine belonging to one of the following categories and have given a written consent to participate in the study.

1. MBBS with Specialisation
2. MBBS
3. Nursing Staff
4. Others

Subjects -

1. Subjects with suspected traumatic brain injury and GCS > 13
2. Of all ages and gender, have understood the study and gave a written informed consent.

Exclusion Criteria:

Subjects -

1. Subjects with active bleeding or scalp laceration
2. Subjects with large extracranial lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-04-25 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the summative usability of CEREBO® | 1 year
  Assessment of ease of use, ease of learning and satisfaction through the questionnaires filled by the operators.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jaimin Shah, Principal Investigator — Civil Hospital India

IPD SHARING:
Plan to Share IPD: No